CLINICAL TRIAL: NCT05754242
Title: Intravenous Vitamin C for the Prevention of Postreperfusion Syndrome in Orthotopic Liver Transplantation From Deceased Donors
Brief Title: Ascorbic Acid to Prevent Postreperfusion Syndrome in Liver Transplantation
Acronym: VITACTOH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Luis Gajate Martín, Principal investigator, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EC 20/606
Record Dates: First submitted 2023-02-15; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Liver Transplantation; Postreperfusion Syndrome; Ascorbic Acid
Keywords: Postreperfusion syndrome
MeSH Terms: interventions — Ascorbic Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascorbic acid (Experimental): 1.5 gr of ascorbic acid diluted in 100 ml of 0.9% saline solution will be administered intravenously during the anhepatic phase of liver transplantation
  Interventions: Drug: Ascorbic acid
- Saline solution (Placebo Comparator): 100 ml of 0.9% saline solution will be administered during the anhepatic phase of liver transplantation
  Interventions: Drug: 0.9% Saline solution

INTERVENTIONS:
Drug: Ascorbic acid — 1.5 gr of ascorbic acid
  Other Names: Vitamin C
  Arms: Ascorbic acid
Drug: 0.9% Saline solution — 100 ml of 0.9% saline solution
  Other Names: Saline
  Arms: Saline solution

SUMMARY:
The goal of this clinical trial is to test the efficacy of intravenous ascorbic acid in preventing the postreperfusion syndrome in liver transplantation. The main questions it aims to answer are:

* Can intravenous ascorbic acid prevent postreperfusion syndrome in liver transplantation ?
* Can ascorbic acid decrease the incidence of liver graft dysfunction after liver transplantation?
* Can ascorbic acid decreased the incidence of postoperative complications after liver transplantation ?

Participants will receive 1.5 g of intravenous ascorbic acid diluted in 100 ml of saline or 100 ml of saline alone, during the anhepatic phase of liver transplantation before reperfusion of the new graft.

Researchers will compared the incidence of postreperfusion syndrome in both groups.

DETAILED DESCRIPTION:
Researches will compared:

* Incidence of postreperfusion syndrome in liver transplantation
* Changes in interleukin values and other inflammatory markers before and after transplantation
* Incidence of liver graft dysfunction between groups
* Incidence of acute renal failure and other complications between groups

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver transplantation

Exclusion Criteria:

* Pregnancy
* Allergy to ascorbic acid
* Nephrolithiasis
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Hyperoxaluria
* Hyperuricemia
* Haemochromatosis
* Sickle cell anemia
* Serum Creatinine > 1.2 mg/dl in women and 1.3 mg/dl in men
* Split liver graft
* Acute liver failure
* Living donor liver transplantation
* Controlled donor asystolia
* Treatment with: indinavir, Vitamin B12, Cyclosporine, iron, deferoxamine, disulfiram

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Postreperfusion syndrome | Within the first 5 minutes after reperfusion of the grafted liver
  When mean arterial pressure decreases by more than 30% relative to the value at the end of the anhepatic phase and lasts for at least 1 min

SECONDARY OUTCOMES:
Ascorbic acid serum levels | Immediately before induction of anesthesia and 12 hours after repercussion of the graft
  Quantification of ascorbic acid levels before and after liver transplantation
Interleukin1beta (IL-1β) levels | Immediately before induction of anesthesia and 12 hours after repercussion of the graft
  Quantification of IL-1β before and after liver transplantation
Tumor Necrosis Factor-alpha (TNFα) levels | Immediately before induction of anesthesia and 12 hours after repercussion of the graft
  Quantification of TNFα before and after liver transplantation
Interleukin-6 levels (IL-6) | Immediately before induction of anesthesia and 12 hours after repercussion of the graft
  Quantification of IL-6 before and after liver transplantation
Interleukin-8 (IL-8) levels | Immediately before induction of anesthesia and 12 hours after repercussion of the graft
  Quantification of IL-8 before and after liver transplantation
Interferon gamma (IFNγ) levels | Immediately before induction of anesthesia and 12 hours after repercussion of the graft
  Quantification of IFNγ before and after liver transplantation
Primary graft dysfunction | First postoperative week
  Incidence of primary graft nonfunction and early graft dysfunction. Graft nonfunction: lack of liver function leading to death if not retransplanted Early graft dysfunction: Olthoff's criteria
Acute renal failure | First postoperative week
  Postoperative renal failure after liver transplantation as Kidney Disease Improving Global Outcomes (KDIGO) definition
Mechanical ventilation | Postoperative until day 30
  Duration of mechanical ventilation (hours) until extubation of the patient
Mortality | Up to day 30
  Mortality of any cause
Length of hospitalization | Through study completion (30 days)
  Length of stay in hospital (days)
Length of Intensive Care Unit (ICU) stay | Through study completion (30 days)
  Length of ICU stay
Duration of vasopressor support after transplantation | Postoperative until study completion (30 days)
  Duration of vasopressor or inotropic support after transplantation
Maximum dose of vasopressor support after transplantation | Postoperative until study completion (30 days)
  Maximum dose of vasopressor or inotropic support after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Luis Gajate, MD PhD, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Hospital Universitario RAmon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication
Access Criteria: Access by mail to principal investigator: gajate.luis@gmail.com

REFERENCES:
- [Background] Aggarwal S, Kang Y, Freeman JA, Fortunato FL, Pinsky MR. Postreperfusion syndrome: cardiovascular collapse following hepatic reperfusion during liver transplantation. Transplant Proc. 1987 Aug;19(4 Suppl 3):54-5. No abstract available. PMID 3303534
- [Background] Siniscalchi A, Dante A, Spedicato S, Riganello L, Zanoni A, Cimatti M, Pierucci E, Bernardi E, Miklosova Z, Moretti C, Faenza S. Hyperdynamic circulation in acute liver failure: reperfusion syndrome and outcome following liver transplantation. Transplant Proc. 2010 May;42(4):1197-9. doi: 10.1016/j.transproceed.2010.03.097. PMID 20534260
- [Background] Paugam-Burtz C, Kavafyan J, Merckx P, Dahmani S, Sommacale D, Ramsay M, Belghiti J, Mantz J. Postreperfusion syndrome during liver transplantation for cirrhosis: outcome and predictors. Liver Transpl. 2009 May;15(5):522-9. doi: 10.1002/lt.21730. PMID 19399736
- [Background] Blanot S, Gillon MC, Lopez I, Ecoffey C. Circulating endotoxins and postreperfusion syndrome during orthotopic liver transplantation. Transplantation. 1995 Jul 15;60(1):103-6. doi: 10.1097/00007890-199507150-00019. No abstract available. PMID 7624932
- [Background] Bezinover D, Kadry Z, McCullough P, McQuillan PM, Uemura T, Welker K, Mastro AM, Janicki PK. Release of cytokines and hemodynamic instability during the reperfusion of a liver graft. Liver Transpl. 2011 Mar;17(3):324-30. doi: 10.1002/lt.22227. PMID 21384515
- [Background] Blanot S, Gillon MC, Ecoffey C, Lopez I. Circulating endotoxins during orthotopic liver transplantation and post-reperfusion syndrome. Lancet. 1993 Oct 2;342(8875):859-60. doi: 10.1016/0140-6736(93)92715-6. No abstract available. PMID 8104281
- [Background] Ishine N, Yagi T, Ishikawa T, Sasaki H, Nakagawa K, Tanaka N. Hemodynamic analysis of post-reperfusion syndrome and the effect of preventing this syndrome using thromboxane A2 synthetase inhibitor (OKY-046) in swine liver transplantation. Transplant Proc. 1997 Feb-Mar;29(1-2):378-81. doi: 10.1016/s0041-1345(96)00127-3. No abstract available. PMID 9123045
- [Background] Girn HR, Ahilathirunayagam S, Mavor AI, Homer-Vanniasinkam S. Reperfusion syndrome: cellular mechanisms of microvascular dysfunction and potential therapeutic strategies. Vasc Endovascular Surg. 2007 Aug-Sep;41(4):277-93. doi: 10.1177/1538574407304510. PMID 17704330
- [Background] Wilson JX. Mechanism of action of vitamin C in sepsis: ascorbate modulates redox signaling in endothelium. Biofactors. 2009 Jan-Feb;35(1):5-13. doi: 10.1002/biof.7. PMID 19319840
- [Background] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036
- [Background] Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's requirement in septic shock. J Res Pharm Pract. 2016 Apr-Jun;5(2):94-100. doi: 10.4103/2279-042X.179569. PMID 27162802
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Derived] Gajate L, de la Hoz I, Espino M, Martin Gonzalez MDC, Fernandez Martin C, Martin-Grande A, Parise Roux D, Pastor O, Villahoz J, Rodriguez-Gandia MA, Nuno Vazquez J. Intravenous Ascorbic Acid for the Prevention of Postreperfusion Syndrome in Orthotopic Liver Transplantation: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 15;12:e50091. doi: 10.2196/50091. PMID 38100226